CLINICAL TRIAL: NCT03920696
Title: Pityriasis Lichenoides: Anatomo-clinical Aspects and Follow-up Monocentric Retrospective Study
Brief Title: Pityriasis Lichenoides : Anatomo-clinical Aspects and Follow-up
Acronym: EtudePL
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP180538
Record Dates: First submitted 2019-03-12; First posted 2019-04-19 (Actual); Last update posted 2019-04-19 (Actual); Status verified 2019-02

CONDITIONS: Pityriasis Lichenoides
Keywords: Pityriasis Lichenoides;; cutaneous lymphoma; lymphoproliferation
MeSH Terms: conditions — Pityriasis Lichenoides; Lymphoma, T-Cell, Cutaneous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Introduction: Pityriasis lichenoides (PL) is an inflammatory dermatitis of undetermined origin consisting of specific papular lesions reflecting an "indolent" lymphoproliferative state.

The current classification is confusing because it mixes semiological and chronological notions.

The objectives of this study are to better describe the clinical, epidemiological, histological, phenotypic and evolutionary aspects of PL in an adult population.

Methods: Investigators will perform a retrospective cohort study including patients with clinical and histological diagnosis of PL from the coding of the Department of Pathology of Henri-Mondor Hospital and from medical records and photographs of lesions if available, between January 2012 and August 2018. A follow-up telephone interviews will also be proposed to each patient to collect evolution data. Photographs will be systematically reviewed as well as cutaneous samples and a genomic analysis will be performed.

Conclusion: Investigators would like to better understand clinical, histological features and evolutionary aspects of PL in an adult population.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patients with Pityriasis Lichenoides selected from histological coding OT0431, seen at Henri Mondor and with a diagnosis verified from medical records.

Exclusion Criteria:

* Histological coding error
* Histological records of patients in care outside Henri Mondor (cases referred for histological expertise only but not seen clinically)
* Clinical lesions incompatible with Pityriasis Lichenoides according to classically published semiological data
* Missing or insufficient medical records for data exploitation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with Pityriasis Lichenoides
Sampling Method: Non-Probability Sample
Enrollment: 52 (Estimated)
Dates: Start 2019-05-01 (Estimated); Primary Completion 2019-11-01 (Estimated); Study Completion 2019-11-01 (Estimated)

PRIMARY OUTCOMES:
To study clinical Aspects of Pityriasis Lichenoides on a large series of adult patients | It will be measured within 6 months of enrollment
  Epidemiological and and clinical aspect description of the lesions from medical charts and photographs: age, sex, suspected trigger of the disease, past medical history, frequency of necrotic lesions, topography of lesions, fever, altered general conditions, treatment modalities of the flare.

SECONDARY OUTCOMES:
To study histological features of Pityriasis Lichenoides | It will be measured within 6 months of enrollment
  The histological description will make use of a centralized re-reading of the slides according to a standardized grid (appearance of the epidermis, type and topography of the dermal infiltrate, results of the immunolabelings etc ...). The investigators aim to investigate the frequency of patients with patterns of pityriasis lichenoides mimicking lymphomatoid papulosis or mycosis fungoides and to correlate the histological aspect with clinical lesions.
To study molecular features of Pityriasis Lichenoides | It will be measured within 6 months of enrollment
  number of clone T in the skin and in the blood.
To study the treatment during patients' monitoring | It will be measured within 6 months of enrollment
  number of patients with need of a prolonged treatment
To study the duration of outbreak during patients' monitoring | It will be measured within 6 months of enrollment
  the time to healing
To study the relapse during patients' monitoring | It will be measured within 6 months of enrollment
  the number of relapses
To study the number of outbreaks during patients' monitoring | It will be measured within 6 months of enrollment
  the number of outbreaks

CONTACTS AND LOCATIONS:
Overall Officials: Saskia ORO, Doctor, Principal Investigator — Assistance Publique Hôpitaux de Paris - CHU Henri Mondor - Créteil

IPD SHARING:
Plan to Share IPD: No
DATAS ARE OWN BY ASSISTANCE PUBLIQUE - HOPITAUX DE PARIS, PLEASE CONTACT SPONSOR FOR FURTHER INFORMATION

REFERENCES:
- [Background] Bowers S, Warshaw EM. Pityriasis lichenoides and its subtypes. J Am Acad Dermatol. 2006 Oct;55(4):557-72; quiz 573-6. doi: 10.1016/j.jaad.2005.07.058. PMID 17010734
- [Background] Zang JB, Coates SJ, Huang J, Vonderheid EC, Cohen BA. Pityriasis lichenoides: Long-term follow-up study. Pediatr Dermatol. 2018 Mar;35(2):213-219. doi: 10.1111/pde.13396. Epub 2018 Jan 9. PMID 29315771
- [Background] Lalevee S, Ortonne N, Hotz C, Schlemmer F, Beldi-Ferchiou A, Delfau-Larue MH, Wolkenstein P, Chosidow O, Ingen-Housz-Oro S. Febrile ulceronecrotic Mucha Habermann disease mimicking aggressive epidermotropic CD8+ cytotoxic T-cell lymphoma: a diagnostic challenge. Eur J Dermatol. 2018 Dec 1;28(6):834-835. doi: 10.1684/ejd.2018.3410. No abstract available. PMID 30325315
- [Background] Geller L, Antonov NK, Lauren CT, Morel KD, Garzon MC. Pityriasis Lichenoides in Childhood: Review of Clinical Presentation and Treatment Options. Pediatr Dermatol. 2015 Sep-Oct;32(5):579-92. doi: 10.1111/pde.12581. Epub 2015 Mar 26. PMID 25816855
- [Background] Nair PS. A clinical and histopathological study of pityriasis lichenoides. Indian J Dermatol Venereol Leprol. 2007 Mar-Apr;73(2):100-2. doi: 10.4103/0378-6323.31894. PMID 17456915
- [Background] Khachemoune A, Blyumin ML. Pityriasis lichenoides: pathophysiology, classification, and treatment. Am J Clin Dermatol. 2007;8(1):29-36. doi: 10.2165/00128071-200708010-00004. PMID 17298104
- [Background] Zaaroura H, Sahar D, Bick T, Bergman R. Relationship Between Pityriasis Lichenoides and Mycosis Fungoides: A Clinicopathological, Immunohistochemical, and Molecular Study. Am J Dermatopathol. 2018 Jun;40(6):409-415. doi: 10.1097/DAD.0000000000001057. PMID 29210716
- [Background] Sibbald C, Pope E. Systematic review of cases of cutaneous T-cell lymphoma transformation in pityriasis lichenoides and small plaque parapsoriasis. Br J Dermatol. 2016 Oct;175(4):807-9. doi: 10.1111/bjd.14605. Epub 2016 Jun 20. No abstract available. PMID 27031678
- [Background] Vonderheid EC, Kadin ME, Telang GH. Commentary about papular mycosis fungoides, lymphomatoid papulosis and lymphomatoid pityriasis lichenoides: more similarities than differences. J Cutan Pathol. 2016 Apr;43(4):303-12. doi: 10.1111/cup.12653. Epub 2015 Dec 22. No abstract available. PMID 26566599